CLINICAL TRIAL: NCT00255216
Title: Policosanol for the Treatment of Hypercholesterolemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Poli-01
Record Dates: First submitted 2005-11-16; First posted 2005-11-18 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2005-10

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Capsules

INTERVENTIONS:
Drug: Policosanol supplement (oral capsule) vs. placebo

SUMMARY:
Policosanol, a compound derived from sugar cane wax and available in health food stores across the United States, is a popular non-prescription product for treating hypercholesterolemia. Virtually all of the published medical literature on policosanol has been authored by research groups in Cuba.

This study will assess the short-term safety and efficacy of policosanol in healthy adults who have a baseline LDL-C of 130-200. The recruitment population will be derived from primary care clinics consisting primarily of Caucasian and African-American patients. The primary outcome measurements will be the percentage change in LDL-C. Secondary outcomes will include changes in total cholesterol, HDL-C, triglycerides, C-reactive protein, and lipoprotein sub-particles. This will be the first known randomized clinical trial of policosanol in North America.

The data derived from this pilot study regarding the lipid lowering effects of policosanol will be used to support applications for further funding through institutions outside the Carolinas Healthcare System including the National Institute of Health (NIH).

Specific Aim: To independently corroborate the lipid lowering effects of policosanol in a small pilot study.

DETAILED DESCRIPTION:
Policosanol, a compound derived from sugar cane wax and available in health food stores across the United States, is a popular non-prescription product for treating hypercholesterolemia. Policosanol has been used in Cuba since 1991 to treat high cholesterol. Virtually all of the published medical literature on policosanol has been authored by research groups in Cuba. According to the Cuban data, policosanol can lower total cholesterol, lower low-density lipoprotein cholesterol (LDL-C), and raise high-density lipoprotein cholesterol (HDL-C). Based on post-marketing surveys, this drug appears to be devoid of any biochemical, hematological, or clinical adverse effects.

Confirmation of this data on policosanol by scientifically rigorous experiments and trials in this country would provide a safe and effective therapeutic option for the treatment of hypercholesterolemia. Consequently, policosanol has the potential to become a valuable tool in the fight against coronary heart disease - a major cause of mortality in the United States.

This pilot study will assess the short-term safety and efficacy of policosanol in healthy adults who have a baseline LDL-C of 130-200. The recruitment population will be derived from primary care clinics consisting primarily of Caucasian and African-American patients. The primary outcome measurements will be the percentage change in LDL-C. Secondary outcomes will include changes in total cholesterol, HDL-C, triglycerides, C-reactive protein, and lipoprotein sub-particles. This will be the first known randomized clinical trial of policosanol in North America.

The data derived from this pilot study regarding the lipid lowering effects of policosanol will be used to support applications for further funding through institutions outside the Carolinas Healthcare System including the National Institute of Health (NIH). Future studies could include an assessment of the effects of policosanol on other markers for coronary heart disease and potential use in combination with current lipid medications. The overall goal is to perform a large multi-center clinical outcome trial to establish the precise clinical benefits of policosanol.

Summary: Demonstration of the lipid-lowering ability of policosanol is an initial step in providing a safe, cost-effective therapy for hypercholesterolemia, thereby advancing the treatment and prevention of cardiovascular disease in this country.

Specific Aim: To independently corroborate the lipid lowering effects of policosanol in a small pilot study.

Hypotheses: After 8 weeks of therapy policosanol 40 mg/day will:

1. Produce a statistically significant reduction in LDL-C compared to placebo.
2. Provide a statistically significant reduction in LDL particle number and C-reactive protein.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* Males, or females who are not pregnant and have a highly reliable contraception method (i.e. hormonal or surgical contraception)
* Baseline LDL-C between 130 and 200

Exclusion Criteria

* History of Coronary Artery Disease - Patients will be excluded if they have been told at any time that they have heart disease based on a history of abnormal EKG, stress test, or coronary catheterization.
* History of Cerebrovascular Disease - Patients with a history of stroke or TIA will be excluded from the study.
* History of Congestive Heart Disease - Patients will be excluded if they have a history of congestive heart failure, regardless of the underlying cause or stage of disease. This will be true even if patients do not have a history of coronary artery disease.
* History of Diabetes - Patients will be asked if they have ever been diagnosed with any type of diabetes in the past. All patients with diabetes including type I, type II, and gestational diabetes will be excluded.
* History of Renal Impairment - Any patient with a history of kidney problems including transient renal impairment or current renal insufficiency will be excluded.
* History of Uncontrolled Hypertension - If patients report a history of poorly controlled blood pressure, defined as systolic blood pressure consistently over 140 or diastolic blood pressure consistently greater than 90, they will be excluded. Blood pressure will be checked at the beginning of the study and patients will be excluded if the initial reading reveals a systolic blood pressure over 160 and/or a diastolic blood pressure over 100.
* History of Untreated or Clinically Evident Thyroid Disease - Patients will be excluded if they report a history of untreated thyroid disease or current symptoms of an untreated thyroid disorder.
* Currently taking medications or supplements with known or potential lipid-altering effects including: phytosterols, statins, cholestin, niacin, fibrates, psyllium fiber, bile acid sequestrants, diabetic medications, and weight control medications such as orlistat
* Currently having residual side effects from a previously discontinued lipid medication
* Pregnancy or breastfeeding
* Triglycerides > 300 at baseline
* Patients with clinical atherosclerotic disease which would be considered a coronary heart disease risk equivalent per ATP III guidelines - including carotid artery disease, peripheral arterial disease, and abdominal aortic aneurysm.
* Patients with 2 or more cardiac risk factors and over 20% risk of coronary disease according to their 10- year Framingham risk assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-01; Study Completion 2005-08

PRIMARY OUTCOMES:
Primary Outcome Variables:
Percent change in LDL-C between baseline and 8 weeks in the policosanol and placebo arms.

SECONDARY OUTCOMES:
Secondary Outcome Variables:
Percent change between baseline and 8 weeks in both study arms for the following parameters:
• total cholesterol, HDL-C, and triglycerides
• hs-CRP
• LDL Particle concentration
• ALT
• Adverse effects profile

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Dulin, MD PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Center for Cardiovascular Health, Charlotte, North Carolina, United States